CLINICAL TRIAL: NCT03365830
Title: Impact of Reproductive Problems on Physical, Emotional, Social Life Areas in Couples Receiving Infertility Treatment
Brief Title: Impact of Reproductive Problems on Couples
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Murat Dogan, primer investigator, Acibadem University
Other Study IDs: Ob&Gyn Fulya2
Record Dates: First submitted 2017-11-29; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FertQol, Beck's Depression Inventory, Beck's Anxiety Inventory — These 3 scale will be given to patients to fill up who takes infertility treatments

SUMMARY:
Reproduction is in fact the most basic instinct of all living things. The fertility of a woman is both a biological fact and a determinant of gender role in society. Motherhood is still seen as the primary role for women in society. Infertility, which manifests itself as a sudden and unexpected life crisis, is an unexpected, perhaps unexplained, condition that spreads over a long period of time, creates extreme stress and forces adjustment mechanisms. Infertility can affect the quality of life by adversely affecting the physical, emotional, social and relational living spaces of people.

The present study examines the effects of reproductive problems on the quality of life in women who receive infertility treatment, and in the direction of the results obtained, the treatment recipients of the health workers are planned to help develop a holistic perspective that takes into account not only reproductive problems but also other affected living areas.

DETAILED DESCRIPTION:
Infertility is a psychological threat, emotional stress, economically expensive, painful and complex life crisis for the treatment for couples. Infertility has negative effects on social and psychological well-being rather than physical health. Infertile people accept this situation as a serious apology, and as a result of their emotional feeling, they are isolated from their surroundings over time. Therefore, infertility is not a simple gynecologic syndrome, and it is a condition that especially affects the woman very biologically, psychologically and socially, resulting in a decrease in health and quality of life. While infertility is not a life threatening health problem, the couple threatens healthy life with negative effects on mental health and quality of life and is defined as a life crisis by some authors. Studies in infertile couples have shown that women experience more anxiety, depression, stress and hostility in their lives than men, and that sexual life is negatively affected.

Today, unforeseen infertility, often unexplained and unpredictable, is considered to have created a stressful situation that pushes the coping mechanisms for a couple and destroys the sense of health and integrity.

The more a woman's identity is defined by her being a mother, the greater the amount of her psychological distress and disability. The longer the duration of infertility, the more dominance and hopelessness dominate and this can result in a greater depression. Generally, psychosocial effects of infertility also affect the components of quality of life in a negative way. The most affected areas are mental health, emotional behavior, environmental psychology, physical and social functions.

In many studies, it was determined that stress, anxiety and depression scores of infertile couples were higher than the fertile population. Anger, nervousness, decreased self-esteem, poor interpersonal relationships, reduced life satisfaction, anxiety and depression are frequently seen psychological disorders associated with infertility.

As a result, infertility is a stressful event for couples with children, and it is also a condition that affects the relationship of couples. The infertile couples have profoundly affected their marriages and social lives because of the long treatment duration, the destructive effect on the continuing mental health, the complexity of the treatment procedures, the unusual and long steps required and the consequences of the IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of infertility,
2. IVF therapy
3. At least elementary school graduate,
4. Married,
5. Communication is not obstacle,
6. Couples who agree to participate in the work

Exclusion Criteria:

* Other than inclusion criteria

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples who takes IVF treatment
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Cronbach alpha value of emotions, general health, cognitive skills and performance of activities of daily living, partnership, and social and family relationships | 12 months
  The fertility quality of life (FertiQoL) measure specifically evaluates the impact of fertility problems in various life areas. The aim of this study was to examine the relationship between FertiQoL and Beck's Depression Inventory and Beck's Anxiety Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Fulya Hospital, Istanbul, Besiktas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dural O, Yasa C, Keyif B, Celiksoy H, Demiral I, Yuksel Ozgor B, Gungor Ugurlucan F, Bastu E. Effect of infertility on quality of life of women: a validation study of the Turkish FertiQoL. Hum Fertil (Camb). 2016 Sep;19(3):186-91. doi: 10.1080/14647273.2016.1214754. Epub 2016 Aug 2. PMID 27486018
- See also: FertiQol — http://sites.cardiff.ac.uk/fertiqol/